CLINICAL TRIAL: NCT05878249
Title: Role Of Wound Lavage in Direct Pulp Capping Of Permanent Teeth With Carious Exposure: A Randomized Controlled Trial
Brief Title: Role Of Wound Lavage in Direct Pulp Capping Of Permanent Teeth With Carious Exposure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ANSHU SINGH
Record Dates: First submitted 2023-05-05; First posted 2023-05-26 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-05

CONDITIONS: Reversible Pulpitis
MeSH Terms: interventions — Saline Solution; Sodium Hypochlorite; Edetic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- wound lavage with normal saline (Experimental): after removing caries and achieving hemostasis wound lavage of the exposed pulp will be done with 5 ml of Normal saline for 30 seconds
  Interventions: Procedure: wound lavage with normal saline
- wound lavage with sodium hypochlorite (Experimental): after removing caries and achieving hemostasis wound lavage of the exposed pulp will be done with 5 ml of 2.5% sodium hypochlorite (NaOCl) for 30 seconds
  Interventions: Procedure: wound lavage with sodium hypochlorite
- wound lavage with Ethylenediaminetetraacetic acid(EDTA) (Experimental): after removing caries and achieving hemostasis wound lavage of the exposed pulp will be done with 12%Ethylenediaminetetraacetic acid(EDTA) for 5 minutes
  Interventions: Procedure: wound lavage with Ethylenediaminetetraacetic acid(EDTA)
- wound lavage with sodium hypochlorite followed by Ethylenediaminetetraacetic acid (Experimental): after removing caries and achieving hemostasis wound lavage of the exposed pulp will be done with 5 ml of 2.5%sodium hypochlorite (NaOCl) for 30 seconds followed by 12%Ethylenediaminetetraacetic acid(EDTA) for 5 minutes
  Interventions: Procedure: wound lavage with sodium hypochlorite followed by Ethylenediaminetetraacetic acid

INTERVENTIONS:
Procedure: wound lavage with normal saline — After removing caries and achieving hemostasis after removing caries and achieving hemostasis, wound lavage of the exposed pulp will be done with 5 ml of Normal saline for 30 seconds
  Arms: wound lavage with normal saline
Procedure: wound lavage with sodium hypochlorite — after removing caries and achieving hemostasis wound lavage of the exposed pulp will be done with 5 ml of 2.5% sodium hypochlorite (NaOCl) for 30 seconds,Subsequently the cavity will be flushed with saline for 10 s and blotted dry using sterile cotton pellets
  Arms: wound lavage with sodium hypochlorite
Procedure: wound lavage with Ethylenediaminetetraacetic acid(EDTA) — after removing caries and achieving hemostasis wound lavage of the exposed pulp will be done with 12% Ethylenediaminetetraacetic acid for 5minutes ,Subsequently, the cavity will be flushed with saline for 10 s and blotted dry using sterile cotton pellets.
  Arms: wound lavage with Ethylenediaminetetraacetic acid(EDTA)
Procedure: wound lavage with sodium hypochlorite followed by Ethylenediaminetetraacetic acid — fter removing caries and achieving hemostasis wound lavage of the exposed pulp will be done with 5 ml of 2.5%sodium hypochlorite (NaOCl) for 30 seconds followed by 12%Ethylenediaminetetraacetic acid(EDTA) for 5 minutes.Subsequently, the cavity will be flushed with saline for 10 s and blotted dry using sterile cotton pellets.
  Arms: wound lavage with sodium hypochlorite followed by Ethylenediaminetetraacetic acid

SUMMARY:
the purpose of the study is to investigate the outcome of wound lavage agents Sodium hypochlorite and Ethylenediaminetetraacetic acid (EDTA) in direct pulp capping of mature permanent teeth with carious exposure.

DETAILED DESCRIPTION:
With the growth of advanced pulp biology and bioactive materials today, management of deep carious lesions has come to a more conservative approach. Vital pulp therapy (VPT), comprising direct pulp capping, partial pulpotomy, and coronal pulpotomy, has been proposed as an alternative treatment to the traditional root canal treatment. Although there seems to be an agreement on the appropriate pulp dressing materials, the recommended irrigant for VPT in permanent teeth is less studied. Dentin matrix is a reservoir of bioactive molecules that are sequestered during dentinogenesis.The releasable growth factors from dentine provide source of cell signaling molecules for initiating repair and regeneration. Evidence shows that EDTA has ability to release growth factors from dentine matrix and it also promotes cell survival,attachment,growth and differentiation. Sodium hypochlorite has high efficacy against biofilms and its semi selective tissue dissolving properties on necrotic rather than vital soft tissue makes it ideal for dentin/pulp wound lavage.In direct pulp capping ,wound lavage with sodium hypochlorite has shown to reduce postoperative pain and early painful failures. However there is a lack of well designed clinical trials on pulp wound lavage.

The aim of this study is to investigate the outcome of wound lavage agents Sodium hypochlorite and EDTA in direct pulp capping of mature permanent posterior teeth with carious exposure Study will be conducted in Post Graduate Institute of Dental Sciences, Rohtak in department of Conservative Dentistry & Endodontics.Time Frame of the study will be 18 months and Patients of age 18-50 years will be enrolled in this study.

After caries excavation, patients will be randomly allocated into four groups- Group I-normal saline, Group II-sodium hypochlorite, Group III-EDTA, Group IV-Sodium hypochlorite followed by EDTA. Washing of the pulp wound will be done with respective allocated solution and then tooth in both groups will be restored according to standard protocol.

Primary outcome variables recorded will be clinical and radiographic success rates after 6 and 12 months from the treatment.

Secondary outcome measure will be reduction in post operative pain after 7days of the treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient willing to participate in the study.
2. Age group- 18-50 years.
3. Mature permanent mandibular posterior teeth (molars or premolars) with reversible pulpitis.
4. Teeth with extremely deep caries (Caries penetrating entire thickness of dentine) responding within normal limits to the cold test and Electric pulp test.
5. Teeth with normal apical tissues(not showing any rarefaction on the intraoral periapical radiograph)

Exclusion Criteria:

1. Primary teeth.
2. Teeth with irreversible pulpitis (spontaneous pain) or pulp necrosis, chronic periodontitis, cracked tooth, internal or external resorption, calcified canals, associated with sinus tract, and furcation or apical radiolucency.
3. Immuno-compromised, diabetic, pregnant and hypertensive patients.
4. Positive history of antibiotic within past one month and analgesic since one week use of the treatment

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
clinical and radiographic success at 6 and 12 months. | 12 months
  Clinical success criteria-
  * Positive response on cold testing
  * Absence of sign and symptoms of spontaneous pain or pain on stimulus and discomfort.
  * No tenderness to palpation or percussion and the tooth is functional.
  * Normal tooth mobility and no periodontal probing pocket depth.
  * Soft tissues around tooth are normal with no swelling or sinus tract.
  Radiographic success criteria-
  * Absence of any periapical or interradicular radiolucency
  * Absence of internal or external root resorption
  * Periapical Index score < 2 according to Orstavik et al.

SECONDARY OUTCOMES:
To assess postoperative pain . | 7 days
  To assess incidence and intensity of pain postoperatively at every 24 hours till 7 days using Visual analogue Scale of 0 to 10 centimeter line. Score 0 means no pain and Score 10 means maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: ANSHU SINGH, MDS, Principal Investigator — PGIDS ROHTAK
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No